CLINICAL TRIAL: NCT01858831
Title: Single Oral Dose Study of Atovaquone/Proguanil Hydrochloride Combination Tablets and Atovaquone Suspension. - A Single Oral Dose Study to Investigate Pharmacokinetics of Atovaquone and Proguanil From Combination Tablets and Atovaquone From Atovaquone Suspension in Japanese Healthy Males. -
Brief Title: Single Oral Dose Study of Atovaquone/Proguanil Hydrochloride Combination Tablets and Atovaquone Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 116441
Record Dates: First submitted 2012-03-15; First posted 2013-05-21 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Atovaquone; Proguanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atovaquone/proguanil HCL (Experimental): Atovaquone/proguanil HCL
  Interventions: Drug: Atovaquone/proguanil HCL
- Atovaquone 750 mg (Active Comparator): Atovaquone 750 mg
  Interventions: Drug: Atovaquone
- Atovaquone 1500 mg (Active Comparator): Atovaquone 1500 mg
  Interventions: Drug: Atovaquone

INTERVENTIONS:
Drug: Atovaquone/proguanil HCL — Atovaquone/proguanil HCL
  Arms: Atovaquone/proguanil HCL
Drug: Atovaquone — Atovaquone
  Arms: Atovaquone 1500 mg; Atovaquone 750 mg

SUMMARY:
This study will be a single-center, phase I, randomized, open, in fed condition, parallel, single dose study to evaluate the pharmacokinetics and the safety, tolerability of Atovaquone/proguanil combination tablets and atovaquone suspension in Japanese healthy male subjects.

Serial blood samples will be collected for the determination of the plasma concentration of atovaquone, proguanil and cycloguanil after dosing of atovaquone 1000mg/proguanil 400 mg and the plasma atovaquone concentration of atovaquone 750 and 1500 mg. Safety assessments will be performed for each treatment group.

CYP2C19 contribute to proguanil metabolism. CYP2C19 genotype will be determined in atovaquone/proguanil dosing group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as defined as being free from clinically significant illness or disease as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital sign, laboratory tests and ECG.
* Japanese healthy male between 20 and 55 years of age inclusive, at the time of signing the informed consent.
* Body weight => 50 kg and BMI within the range 18.5- 25 kg/m2
* Non-smoker or ex-smoker having ceased smoking for at least 6 months. (inclusive).
* ALT, alkaline phosphatase and bilirubin below the upper limit of normal (ULN)
* Single QTcB< 450 msec.
* Vital sign within the following ranges; Systolic blood pressure: < 90 mmHg or > 140 mmHg, Diastolic blood pressure: < 45 mmHg or > 90 mmHg, Plus rate: < 45 bpm or > 100 bpm, Body temperature: 37.5 C
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive results of syphilis, HBs antigen, HCV antibody, HIV antibody and HTLV-1 antibody at the time of screening.
* History of any cardiac diseases irrespective of with or without symptom.
* An episode of cardiac syncope within one year before screening period.
* History/evidence of clinically significant pulmonary diseases and hyper/hypo-thyroidism.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug screen.
* History of regular alcohol consumption exceeding, on average, 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 350 mL of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening.
* The subject had participated in a clinical study or post-marketing study with an investigational or a non-investigational product during the previous 4 months preceding the administration of study medication of this study.
* The subject had participated in a clinical study or post-marketing study with an investigational or a non-investigational product during the previous 4 months preceding the administration of study medication of this study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of alcohol, prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy excluding pollen allergy without current symptoms.
* Where participation in the study would result in donation of blood or blood products in excess of 400 mL within a 4 month or 200 mL within 2 month.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
plasma atovaquone concentration | pre, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 120, 168, 216, 336 post dose
plasma proguanil concentration | pre, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 120, 168, 216, 336 post dose
plasma cycloguanil concentration | pre, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 120, 168, 216, 336 post dose

SECONDARY OUTCOMES:
Number of participants with adverse events | up to 336h post dose
Change in Systolic Blood Pressure | at pre-dose, 4, 24, 72, 168 and 336 h post-dose
  Change values at 4, 24, 72, 168 and 336 h post-dose from baseline (pre-dose)
Change in ECG findings | at pre-dose, 4, 72, 168 and 336 h post-dose
  Change at 4, 72, 168 and 336 h post-dose from baseline (pre-dose)
Laboratory | at pre-dose, 72, 168 and 336 h post-dose
  Change values at 72, 168 and 336 h post-dose from baseline (pre-dose)
Change in Diastolic Blood Pressure | at pre-dose, 4, 24, 72, 168 and 336 h post-dose
  Change values at 4, 24, 72, 168 and 336 h post-dose from baseline (pre-dose)
Change in Heart rate | at pre-dose, 4, 24, 72, 168 and 336 h post-dose
  Change values at 4, 24, 72, 168 and 336 h post-dose from baseline (pre-dose)
Change in Hematology values | at pre-dose, 72, 168 and 336 h post-dose
  Change values at 72, 168 and 336 h post-dose from baseline (pre-dose)
Change in Biochemistry values | at pre-dose, 72, 168 and 336 h post-dose
  Change values at 72, 168 and 336 h post-dose from baseline (pre-dose)
Change in Urinalysis values | at pre-dose, 72, 168 and 336 h post-dose
  Change values at 72, 168 and 336 h post-dose from baseline (pre-dose)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kagoshima, Japan

REFERENCES:
- See also: Results for study 116441 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116441?search=study&#rs